CLINICAL TRIAL: NCT01231373
Title: A Randomized, Blinded, Multicenter Study to Evaluate the Efficacy and Safety of Varisolve Polidocanol Endovenous Microfoam (PEM) 0.5% and 1% Compared to Vehicle for the Treatment on Saphenofemoral Junction (SFJ) Incompetence "VANISH-2"
Brief Title: Polidocanol Endovenous Microfoam (PEM) Versus Vehicle for the Treatment of Saphenofemoral Junction (SFJ) Incompetence
Acronym: VANISH-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VAP.VV016
Record Dates: First submitted 2010-10-22; First posted 2010-11-01 (Estimated); Results first posted 2014-04-02 (Estimated); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Varicose Veins
Keywords: varicose veins
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- polidocanol injectable foam, 0.125% (Experimental)
  Interventions: Drug: polidocanol injectable foam, 0.125%
- polidocanol injectable foam, 0.5% (Experimental)
  Interventions: Drug: polidocanol injectable foam, 0.5%
- polidocanol injectable foam, 1.0% (Experimental)
  Interventions: Drug: polidocanol injectable foam, 1.0%
- Vehicle (Placebo Comparator)
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: polidocanol injectable foam, 0.125% — active placebo for blinding
  Arms: polidocanol injectable foam, 0.125%
Drug: polidocanol injectable foam, 0.5% — 0.5% polidocanol foam injection
  Arms: polidocanol injectable foam, 0.5%
Drug: polidocanol injectable foam, 1.0% — 1.0% polidocanol foam injection
  Arms: polidocanol injectable foam, 1.0%
Drug: Vehicle — injection of vehicle comparator
  Arms: Vehicle

SUMMARY:
Varicose veins are enlarged, noticeably bulging veins, which commonly occur in the legs and may cause discomfort. In this study, patients with varicose veins in the legs will be participating. The purpose of this research study is to evaluate the safety and effectiveness of three different concentrations of an investigational drug, Polidocanol Endovenous Microfoam (PEM) compared to vehicle (inactive solution) in treating the symptoms and appearance of varicose veins.

ELIGIBILITY:
Inclusion Criteria:

* Incompetence of SFJ associated with incompetence of the GSV or other major accessory vein
* Ability to comprehend and sign an informed consent document and complete study questionnaires in English
* Ability to record symptoms in accordance with the protocol
* Symptomatic varicose veins
* Visible varicose veins

Exclusion Criteria:

* Patients who only have telangiectatic or reticular veins (Clinical Finding C1, as assessed by CEAP Classification of Venous Disorders).
* Leg obesity impairing the ability to access the vein to be treated and/or to apply post-procedure compression bandaging and stockings
* Ultrasonographic or other evidence of current or previous deep vein thrombosis or occlusion
* Deep vein reflux unless clinically insignificant in comparison to superficial reflux
* Peripheral arterial disease precluding the wearing of post-procedure compression bandaging and stockings
* Reduced mobility
* Major surgery, prolonged hospitalization or pregnancy within 3 months of screening
* Major co-existing disease (e.g. malignancy; pulmonary disease; renal or hepatic insufficiency; serious skin disease/condition that may compromise the ability of the patient to comply with the compression protocol, etc.)
* Known allergic response to polidocanol or heparin, including history of heparin-induced thrombocytopenia, and/or multiple allergic reactions
* Current alcohol or drug abuse
* Pregnant or lactating women
* Women of childbearing potential not using effective contraception
* History of DVT, pulmonary embolism, or stroke

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2010-11; Primary Completion 2011-09 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Dothan, Alabama
  - San Diego, California
  - Lafayette, Indiana
  - Frederick, Maryland
  - Hunt Valley, Maryland
  - Los Alamos, New Mexico
  - Oklahoma City, Oklahoma
  - Monroeville, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Greenville, South Carolina
  - Bellevue, Washington

REFERENCES:
- [Derived] Todd KL 3rd, Wright DI; VANISH-2 Investigator Group. Durability of treatment effect with polidocanol endovenous microfoam on varicose vein symptoms and appearance (VANISH-2). J Vasc Surg Venous Lymphat Disord. 2015 Jul;3(3):258-264.e1. doi: 10.1016/j.jvsv.2015.03.003. Epub 2015 May 6. PMID 26992303

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three (3) patients were randomized but never treated.
Groups:
- Polidocanol Injectable Foam, 0.125%: active placebo for blinding of therapeutic polidocanol dose
- Polidocanol Injectable Foam, 0.5%: lower experimental polidocanol dose
Period: Overall Study
Arm/Group | Vehicle | Polidocanol Injectable Foam, 0.125% | Polidocanol Injectable Foam, 0.5% | Polidocanol Injectable Foam, 1.0%
Started | 59 | 58 | 60 | 58
Patients Receiving Blinded Treatment | 57 | 57 | 60 | 58
Completed | 56 | 57 | 60 | 57
Not Completed | 3 | 1 | 0 | 1
Not completed — Withdrew consent prior to randomization | 2 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Withdrew Consent | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients receiving blinded treatment
Groups:
- Polidocanol Injectable Foam, 0.125%: polidocanol injectable foam active placebo
- Polidocanol Injectable Foam, 0.5%: polidocanol injectable foam lower experimental dose
- Polidocanol Injectable Foam, 1.0%: polidocanol injectable foam therapeutic dose
- Total: Total of all reporting groups
Arm/Group | Vehicle | Polidocanol Injectable Foam, 0.125% | Polidocanol Injectable Foam, 0.5% | Polidocanol Injectable Foam, 1.0% | Total
Number analyzed (Participants) | 57 | 57 | 60 | 58 | 232
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.8 (10.44) | 52.8 (10.06) | 50.4 (9.89) | 50.4 (11.42) | 50.8 (10.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 43 | 40 | 44 | 169
  Male | 15 | 14 | 20 | 14 | 63
Race/Ethnicity, Customized [Number; unit: participants]
  White | 54 | 53 | 55 | 53 | 215
  Black | 2 | 1 | 3 | 0 | 6
  Asian | 0 | 1 | 0 | 1 | 2
  American Indian/Eskimo | 0 | 0 | 0 | 1 | 1
  Other | 1 | 2 | 2 | 3 | 8
Weight [Mean (Standard Deviation); unit: kilograms] | 83.0 (20.22) | 85.3 (16.41) | 88.8 (22.66) | 81.4 (20.22) | 84.8 (20.11)
Height [Mean (Standard Deviation); unit: centimeters] | 169.7 (9.45) | 168.6 (9.38) | 169.6 (10.47) | 169.1 (9.27) | 169.3 (9.61)
Calculated BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.8 (5.76) | 30.1 (19.48) | 30.7 (6.28) | 28.4 (6.45) | 29.5 (6.03)

OUTCOME MEASURES:

1. Primary Outcome: Change in Patient-Reported Symptoms of Varicose Veins (VVSymQ Score)
Description: The 9 varicose vein symptoms were to be assessed and graded on a 6-point (i.e., 0-5) duration scale and an 11-point (i.e., 0-10) intensity scale, and the patient's level activity for that day was to be assessed and graded on the 6-point (i.e., 0-5) duration scale. The 9 varicose vein symptoms assessed using the e-diary were derived from the first question of the modified Venous Insufficiency Epidemiologic and Economic Study-Quality of Life/Symptoms (VEINES-QOL/Sym) instrument. The VVSymQ is a subset of 5 VEINES QOL/Sym items that have been determined in earlier studies to be most important to patients. The daily VVSymQ score is the sum of the duration scores for these 5 symptoms (scores range from 0 to 25). At Visit 2/baseline, Week 8, scores were calculated.
Time Frame: 8 weeks
Population: Number of subjects with a baseline value (VVSymQ) and value at the 8 week visit.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Polidocanol Injectable Foam, 0.5%: experimental dose polidocanol injectable foam, 0.5%
- Polidocanol Injectable Foam, 1.0%: polidocanol injectable foam, 1.0%: Injection of mid-dose PEM
Arm/Group | Vehicle | Polidocanol Injectable Foam, 0.125% | Polidocanol Injectable Foam, 0.5% | Polidocanol Injectable Foam, 1.0%
Number analyzed (Participants) | 54 | 54 | 60 | 57
units on a scale | -2.00 (0.474) | -5.34 (0.476) | -6.01 (0.454) | -5.06 (0.463)
Statistical Analysis 1: Comparison: Vehicle vs Polidocanol Injectable Foam, 0.125%; Comparison of polidocanol treatment groups versus placebo (absolute change from baseline to week 8 in patient assessment of symptoms of varicose veins (VVSymQ) score; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -3.34, 95% CI 2-sided [-4.63 to -2.04]
Statistical Analysis 2: Comparison: Vehicle vs Polidocanol Injectable Foam, 0.5%; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -4.00, 95% CI 2-sided [-5.26 to -2.74]
Statistical Analysis 3: Comparison: Vehicle vs Polidocanol Injectable Foam, 1.0%; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -3.05, 95% CI 2-sided [-4.33 to -1.77]

2. Secondary Outcome: Change From Baseline to 8 Weeks in Appearance as Rated by Patient (PA-V3)
Description: The Patient Self-assessment of Visible Varicose Veins (PA-V3) instrument is a 5-point scale used by patients to evaluate the appearance of their visible varicose veins. On this single-item paper questionnaire, the instructions included a diagram fo the medial view of a leg with the area between the ankle and the groin circled. The patient was instructed to choose 1 of 5 response options that best described the appearance of the visible varicose veins of the leg that was treated in the study. The patient was instructed not to consider the appearance of the leg outside the circled area or of any spider veins. Possible responses ranged from "Not at all noticeable" (a score of 0) to "Extremely noticeable" (a score of 4).
Time Frame: 8 weeks
Population: patients with a baseline and week 8 visit.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Polidocanol Injectable Foam, 1.0%: polidocanol injectable foam, experimental dose 1.0%
Arm/Group | Vehicle | Polidocanol Injectable Foam, 0.125% | Polidocanol Injectable Foam, 0.5% | Polidocanol Injectable Foam, 1.0%
Number analyzed (Participants) | 56 | 56 | 60 | 57
units on a scale | -0.07 (0.080) | -0.74 (0.081) | -0.89 (0.078) | -0.83 (0.080)
Statistical Analysis 1: Comparison: Vehicle vs Polidocanol Injectable Foam, 0.125%; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.66, 95% CI 2-sided [-0.88 to -0.45], Standard Error of Mean 0.081
Statistical Analysis 2: Comparison: Vehicle vs Polidocanol Injectable Foam, 0.5%; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.82, 95% CI 2-sided [-1.04 to -0.61], Standard Error of Mean 0.078
Statistical Analysis 3: Comparison: Vehicle vs Polidocanol Injectable Foam, 1.0%; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.75, 95% CI 2-sided [-0.97 to -0.54]

3. Secondary Outcome: Change From Baseline at 8 Weeks Post-Treatment in IPR-V3 Score--Physician Photographic Review of Appearance
Description: The Independent Photography Review--Visible Varicose Veins (IPR-V3) instrument is a 5-point scale used to assess the appearance of a patient's visible varicose veins. At baseline and Week 8, standardized digital photographs were taken of the medial view of the patient's target leg, from groin to ankle. An independent photography review panel, consisting of 3 trained, blinded clinicians, evaluated the appearance of the patient's visible varicose veins using the IPR-V3 instrument's 5-point scale (0-4, where 0=none and 4=very severe visible varicose veins).
Time Frame: 8 weeks
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Polidocanol Injectable Foam, 1.0%: polidocanol injectable foam, 1.0% experimental dose
Arm/Group | Vehicle | Polidocanol Injectable Foam, 0.125% | Polidocanol Injectable Foam, 0.5% | Polidocanol Injectable Foam, 1.0%
Number analyzed (Participants) | 56 | 57 | 60 | 57
units on a scale | -0.32 (0.133) | -1.55 (0.131) | -1.86 (0.129) | -1.79 (0.130)
Statistical Analysis 1: Comparison: Vehicle vs Polidocanol Injectable Foam, 0.125%; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -1.23, 95% CI 2-sided [-1.59 to -0.87], Standard Error of Mean 0.131
Statistical Analysis 2: Comparison: Vehicle vs Polidocanol Injectable Foam, 0.5%; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -1.54, 95% CI 2-sided [-1.90 to -1.18], Standard Error of Mean 0.129
Statistical Analysis 3: Comparison: Vehicle vs Polidocanol Injectable Foam, 1.0%; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -1.47, 95% CI 2-sided [-1.83 to -1.11], Standard Error of Mean 0.130

ADVERSE EVENTS:
Time Frame: Adverse events that occurred after patient provided informed consent through Visit 5/Week 8 (or Visit 8 for patients receiving open-label PEM 1.0%)
Groups:
- Polidocanol Injectable Foam, 0.125%: polidocanol injectable foam, 0.125% active placebo
- Polidocanol Injectable Foam, 0.5%: polidocanol injectable foam, 0.5% lower experimental dose
- Polidocanol Injectable Foam, 1.0%: polidocanol injectable foam target therapeutic dose
Arm/Group | Vehicle | Polidocanol Injectable Foam, 0.125% | Polidocanol Injectable Foam, 0.5% | Polidocanol Injectable Foam, 1.0%
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/58 | 0/60 | 0/58
Other Adverse Events (participants affected / at risk) | 11/59 | 24/58 | 27/60 | 47/58
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle (N=59) | Polidocanol Injectable Foam, 0.125% (N=58) | Polidocanol Injectable Foam, 0.5% (N=60) | Polidocanol Injectable Foam, 1.0% (N=58)
Infusion site thrombosis (General disorders) | 0 (0) | 6 (6) | 7 (7) | 16 (16)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (7) | 9 (9) | 4 (4) | 10 (10)
Thrombophlebitis superficial (Vascular disorders) | 1 (1) | 4 (4) | 8 (8) | 2 (2)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 2 (2) | 2 (2) | 4 (4)
Hematoma (Vascular disorders) | 1 (1) | 2 (2) | 3 (3) | 3 (3)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 2 (2) | 3 (3)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Tenderness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days